CLINICAL TRIAL: NCT04553809
Title: The Efficacy of Combining Endoscopic Modalities for the Diagnosis of Solitary Pulmonary Lesions
Brief Title: Navigation Endobronchial Ultrasound
Acronym: NEBULA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amanda Dandanell Juul (Other)
Responsible Party: Sponsor-Investigator, Amanda Dandanell Juul, MD, PhD student, University of Southern Denmark
Organization: University of Southern Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ENBPhD
Record Dates: First submitted 2020-09-03; First posted 2020-09-17 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer
Keywords: lung cancer diagnotics
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kontrol (Active Comparator): Patients undergoing examination for lung cancer with the use of electromagnetic navigation bronchoscopy for biopsy sampling
  Interventions: Procedure: ENB
- Intervention (Experimental): Patients undergoing examination for lunge cancer with the use of electromagnetic navigation bronchoscopy and radial endobronchial ultrasound for biopsy sampling.
  Interventions: Procedure: ENB in combination with rEBUS

INTERVENTIONS:
Procedure: ENB — ENB for biopsy sampling of peripheral lung lesion
  Arms: Kontrol
Procedure: ENB in combination with rEBUS — The combination of ENB and rEBUS for biopsy sampling of peripheral lung lesions
  Arms: Intervention

SUMMARY:
Lung cancer is the primary cause of cancer related deaths in Denmark. In order to improve the prognosis diagnosis in earlier stages are needed. This will however require improved sampling techniques from very small lung lesions.

One method involves the use of a radial ultrasound probe inserted in the working channel of the bronchoscope, to more accurately identify the lung lesions before sampling them (rEBUS). The other method involves the use of electromagnetic navigation bronchoscopy (ENB) to guide the operator to the lung lesion.

This study aims to determine whether a combination of rEBUS and ENB is superior to ENB alone in biopsy sampling. The study will be conducted as a non-blinded RCT. Furthermore, we will make an estimate of the hospital costs of the entire diagnostic work up for lung cancer when combining ENB and rEBUS compared to ENB alone.

DETAILED DESCRIPTION:
Background:

Despite recent years' improvement regarding the treatment of lung cancer, it remains the leading cause of cancer deaths in Denmark. This is partly due to many patients being diagnosed in an advanced stage limiting the possibilities of curative treatment. Much attention has therefore been aimed at developing tools for early identification of patients with possible lung cancer . Screening or easy access to CT of the chest may help to identify patients with possible early stage lung cancer. Performing biopsies of small lung lesions in a safe manner without inexpedient complications, however, is an ongoing diagnostic challenge especially for the increasing elderly patient population and patients with decreased lung function. If patients are to benefit from an improved identification of possible early stage lung cancer, it is necessary to also further improve the methods for obtaining biopsies in this patient population in order to decrease the morbidity during the diagnostic work-up and to prepare the patients for treatment in a secure manner.

Current methods for performing biopsies of small lung lesions are transthoracic, endoscopic or surgical. When compared to surgery, the endoscopic methods have the advantages of being easily accessible, cheap, safe with a very low risk of complications, and have limited patient discomfort following the procedure. The major drawback is the diagnostic yield still being significantly lower than surgery.

In recent years, two methods have been developed which seem to improve the diagnostic yield of bronchoscopy for diagnosing peripheral lung lesions. The rationale behind both techniques is to improve identification of the lung lesions prior to performing the biopsies and thereby improving the chance of obtaining representative tissue samples. One method involves the use of a radial ultrasound probe inserted in the working channel of the bronchoscope, which enables the proceduralist to perform radial endobronchial ultrasound (rEBUS) to more accurately identify the lung lesions before sampling them. The other method involves the use of electromagnetic navigation bronchoscopy (ENB) to guide the operator to the lung lesion. One small randomised clinical trial has indicated that the diagnostic yield can be further improved by a multimodal approach, which combines both rEBUS and ENB in the same procedure. The drawbacks of such a combination are however increased costs and procedure time, thus limiting the number of procedures which can be performed within a given time frame.

This PhD thesis aims to determine whether a combination of rEBUS and ENB is superior to ENB alone in patients with suspected lung cancer due to a peripheral lung lesion as well as an estimate of the hospital costs of the entire diagnostic work up for lung cancer when combining ENB and rEBUS as compared to ENB alone.

Hypotheses:

1. The diagnostic yield of ENB in combination with rEBUS is equal to ENB alone in patients with peripheral lung lesions or solitary lung nodules (null hypothesis)
2. The hospital costs of the entire diagnostic work up for lung cancer when combining ENB and rEBUS is the same when compared to an approach with ENB alone (null hypothesis)

Research questions:

1. Is the diagnostic yield of ENB in combination with rEBUS different from ENB alone in diagnosing lung lesions?
2. What are the hospital costs of the entire diagnostic workup for lung cancer when combining ENB and rEBUS in comparing with ENB alone?

Navigation EndoBronchial ULtrAsound (NEBULA):

Hypotheses The study examines the following null-hypothesis: The diagnostic yield of ENB in combination with rEBUS is not superior to ENB alone in patients with peripheral lung lesions or solitary lung nodules.

Objectives To determine which bronchoscopy approach should be considered standard for examining patients with suspected lung cancer due to a peripheral lung lesion.

Methods Study design Multicentre, randomized, non-blinded clinical trial Pre- and post-procedure Preparations prior and following the bronchoscopy procedure are done in accordance with local guidelines. Procedures will be performed either under conscious sedation using midazolam and fentanyl or in general anesthetic depending on the set up of the center performing the procedures. Other medication given during the procedure is also given accordance with local guidelines.

Reference test Histology or cytology results will be used as the reference test for all malignant as well as non-malignant conditions that could be diagnosed based on these. Clinical follow-up including imaging for at least 6 months with no signs of malignancy and results of additional diagnostic procedures will be used as the reference test in patients in which a final diagnosis cannot be established based on histology or cytology results.

Sample size and statistics In a previous study by Eberhardt et al. the diagnostic yield of ENB and combined rEBUS/ENB was 59 % and 88 %, respectively. The diagnostic yield of the intervention arm in the planned study may be lower due to selection of patients with smaller lesions and multicentre approach rather than a single centre study performed by experts. If the total diagnostic yield is 60 % in the control group (ENB) and 80 % in the intervention group (rEBUS/ENB), then a power of 80 % at the 5 % level is obtained with a sample size of 184 patients. Allowing for a 10 % dropout it is planned to enroll 200 patients in the study. The χ2 test, alternatively the Fischer exact test will be used to establish whether there is a difference in the primary endpoint. All results will be assessed using intention to treat principles.

Ethics:

The studies and analyses will be conducted in accordance with the amended Declaration of Helsinki and Data Protection Agency in Denmark and the Medical Ethics Committee.:

The studies do not interfere with choice of other diagnostic tests performed in the patients (e.g. EBUS / EUS-b for mediastinal staging). The patients are treated and followed up according to national and institutional guidelines. The protocols for studies II and III do not influence treatment or follow-up.

Clinical relevance:

The results will help to clarify how one of the most important diagnostic procedures for patients with suspected lung cancer due to a peripheral lung lesion should be used in clinical practice. The results of the project can be directly implemented at a national scale once the results are available.

Economy:

Project expenses are expected to be partially covered by funds from the Kræftens Bekæmpelse - Centre for Lung Cancer Research with a grant of 1 mill. DKK. Funding of expenses for procedures (e.g. scans and invasive procedures) will be covered as part of the lung cancer diagnostic work up "package" covered by the department.

Participating departments:

Currently the following departments have agreed to participate:

* Department of Respiratory Medicine, Bispebjerg Hospital
* Department of Respiratory Medicine, Aalborg University Hospital
* Department of Respiratory Medicine, Odense University Hospital

ELIGIBILITY:
Inclusion Criteria:

* Examination for lung cancer
* Peripheral lung lesion or lung nodule surrounded by normal lung parenchyma
* Written and orally informed consent

Exclusion Criteria:

* Patient has medical devices in which ENB is contraindicated (e.g. implanted pacemaker or defibrillator)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Total diagnostic yield | 6 months
  Total diagnostic yield, being defined as a tissue biopsy allowing a definite diagnosis of either a malignant or benign condition in the lung in proportion to the total number of procedures performed.

SECONDARY OUTCOMES:
Malignant diagnostic yield | 6 months
  Diagnostic yield of malignant conditions, being defined as a tissue biopsy allowing a definite diagnosis of a malignant condition in the lung
Non-malignant diagnostic yield | 6 months
  Diagnostic yield of non-malignant conditions, being defined as a tissue biopsy allowing a definite diagnosis of a benign condition in the lung
Complications | 1 week
  Total proportion of patients with procedure complications
Severe complications | 1 week
  Total proportion of patients with severe procedure complications
Ready to treat | 7 months
  Time from referral to "ready to treat"
Discomfort | 2 weeks
  Patient reported procedure discomfort during the endoscopic procedure. Reported in a questionnaire efter the procedure.
Patient satisfaction | 2 weeks
  Patient reported procedure satisfaction. Reported in a questionnaire after the procedure in a scale from 1 -10.
Procedure time | 1 week
  Procedure time differens between the two arms
Procedure costs | 2 years
  Differens in procedure cost for the two arms, reported in daniske kroner or converted to euro for publications
Entire work-up costs | 2 years
  Hospital costs of the entire diagnostic workup incl. admissions and expenses for treating adverse events from referral to end of "cancer package". Reported in danish kroner or converted to euro for publication.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Dandanell Juul, MD, Principal Investigator — Dept. of Respiratory Medicine, Odense University Hospital
Locations (1):
- Departement of respiratory medicin, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eberhardt R, Anantham D, Ernst A, Feller-Kopman D, Herth F. Multimodality bronchoscopic diagnosis of peripheral lung lesions: a randomized controlled trial. Am J Respir Crit Care Med. 2007 Jul 1;176(1):36-41. doi: 10.1164/rccm.200612-1866OC. Epub 2007 Mar 22. PMID 17379850
- [Background] Brownback KR, Quijano F, Latham HE, Simpson SQ. Electromagnetic navigational bronchoscopy in the diagnosis of lung lesions. J Bronchology Interv Pulmonol. 2012 Apr;19(2):91-7. doi: 10.1097/LBR.0b013e31824dd9a1. PMID 23207349
- [Background] Zhang W, Chen S, Dong X, Lei P. Meta-analysis of the diagnostic yield and safety of electromagnetic navigation bronchoscopy for lung nodules. J Thorac Dis. 2015 May;7(5):799-809. doi: 10.3978/j.issn.2072-1439.2015.04.46. PMID 26101635
- [Background] Ali MS, Trick W, Mba BI, Mohananey D, Sethi J, Musani AI. Radial endobronchial ultrasound for the diagnosis of peripheral pulmonary lesions: A systematic review and meta-analysis. Respirology. 2017 Apr;22(3):443-453. doi: 10.1111/resp.12980. Epub 2017 Feb 8. PMID 28177181
- [Background] Khan KA, Nardelli P, Jaeger A, O'Shea C, Cantillon-Murphy P, Kennedy MP. Navigational Bronchoscopy for Early Lung Cancer: A Road to Therapy. Adv Ther. 2016 Apr;33(4):580-96. doi: 10.1007/s12325-016-0319-4. Epub 2016 Mar 22. PMID 27084723
- [Background] Herth FJ, Eberhardt R, Becker HD, Ernst A. Endobronchial ultrasound-guided transbronchial lung biopsy in fluoroscopically invisible solitary pulmonary nodules: a prospective trial. Chest. 2006 Jan;129(1):147-50. doi: 10.1378/chest.129.1.147. PMID 16424425
- [Background] Wang Memoli JS, Nietert PJ, Silvestri GA. Meta-analysis of guided bronchoscopy for the evaluation of the pulmonary nodule. Chest. 2012 Aug;142(2):385-393. doi: 10.1378/chest.11-1764. PMID 21980059
- [Background] Haas AR, Vachani A, Sterman DH. Advances in diagnostic bronchoscopy. Am J Respir Crit Care Med. 2010 Sep 1;182(5):589-97. doi: 10.1164/rccm.201002-0186CI. Epub 2010 Apr 8. PMID 20378726
- [Background] Munoz-Largacha JA, Litle VR, Fernando HC. Navigation bronchoscopy for diagnosis and small nodule location. J Thorac Dis. 2017 Mar;9(Suppl 2):S98-S103. doi: 10.21037/jtd.2017.01.57. PMID 28446971
- [Background] Evison M, Crosbie PA, Morris J, Martin J, Barber PV, Booton R. Can computed tomography characteristics predict outcomes in patients undergoing radial endobronchial ultrasound-guided biopsy of peripheral lung lesions? J Thorac Oncol. 2014 Sep;9(9):1393-7. doi: 10.1097/JTO.0000000000000249. PMID 25122434
- [Background] Schreiber G, McCrory DC. Performance characteristics of different modalities for diagnosis of suspected lung cancer: summary of published evidence. Chest. 2003 Jan;123(1 Suppl):115S-128S. doi: 10.1378/chest.123.1_suppl.115s. PMID 12527571
- See also: Technology Assessment Unit of the McGill University Health Centre (MUHC): — https://muhc.ca/sites/default/files/micro/m-TAU/muhc_tau_2016_74_ebus_enb.pdf